CLINICAL TRIAL: NCT04695639
Title: Correlation Between Selective Motor Control and Upper Extremity Functions in Children With Hemiparetic Cerebral Palsy
Brief Title: Selective Motor Control and Upper Extremity Functions in Children With Hemiparetic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira M Abd-elmonem, PHD, principle investigator, Cairo University
Other Study IDs: Selective Motor Control
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
Keywords: Cerebral pals; selective voluntary motor control; upper extremity function; hand grip strength
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort group: A convenient sample of children with spastic hemiparetic CP of both genders will participate in this study. To avoid type II error, sample size calculation was performed prior to the study, based on data of pilot study, using G*POWER statistical software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) [Exact tests- correlational study, α=0.05, β=0.2, and effect size = 0.4] and revealed that the appropriate sample size for this study is N=46.
  Interventions: Other: Test of Arm Selective Control; Other: Hand Held Dynamometer; Other: Quality of Upper Extremity Skill Test

INTERVENTIONS:
Other: Test of Arm Selective Control — It will be used to assess selective voluntary motor control. It is a reliable and valid evaluation tool used to quantify and describe selective voluntary motor control in children with spastic cerebral palsy. The goal of the assessment is to systematically evaluate a person's ability to move the upper extremity with selective voluntary motor control by observing movement control, coordination, fluency, mirroring, and speed at each joint, and then assigning a grade, all in 'real time. Clinically this measure may guide the selection of medical, surgical, or therapy interventions and may improve outcome prognosis after brief training. Raters demonstrated excellent reliability in assessing upper extremity SVMC in a group of children with hemiplegic, diplegic, and quadriplegic CP using the Ttest of arm selective control
Other: Hand Held Dynamometer — Hand held dynamometer (Camry Digital Hand Dynamometer Grip Strength, Model EH101-37, China) will be used to assess hand grip strength of the affected upper extremity. It is generally small, portable and relatively cheap reliable measurement instruments to measure muscle strength of the arm and hand in children with spastic cerebral pasly. It is used to measure strength; maximal voluntary isometric contraction; objectively in kilograms, pounds or newtons. Such devices have been proven to have good to excellent reliability in different populations. It represents an easily accessible way to assess muscle weakness in children with cerebral palsy and the overall reliability is considered to be good.
Other: Quality of Upper Extremity Skill Test — It will be used to assess function of the affected upper extremity. It is a reliable and valid outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. It is designed to be used with children who have neuromotor dysfunction with spasticity and has been validated with children from 18 months to 8 years of age.

SUMMARY:
Identification of musculoskeletal and neuromuscular factors that affect the integrity and functional performance in children with cerebral palsy is very essential as it enables multidisciplinary rehabilitation team to design the proper intervention to improve functional performance and independence for those children.

DETAILED DESCRIPTION:
Limited literature is available regarding the relation between selective voluntary motor control and motor functions in children with cerebral palsy. Up to our knowledge this is the first study intending to investigate the influence of selective voluntary motor control on upper extremity function in children with spastic cerebral palsy. Therefore, the current study will be conducted to investigate the correlation between selective voluntary motor control and upper extremity functions in children with spastic hemiparetic cerebral palsy.

It is hypothesized that:-

1. There is no relation between SVMC and upper limb function in children with spastic hemiparetic CP.
2. There is no relation between upper extremity SVMC and hand grip strength in children with spastic hemiparetic CP.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 4 to 8 years.
* Both genders.
* Diagnosis of spastic hemiparetic cerebral palsy.
* Level I-IV on Manual Ability Classification System.
* Spasticity grade 1 to 2 on Modified Ashworth Scale.
* Level I-III on Gross Motor Classification System .

Exclusion Criteria:

* Significant mental or psychological problems.
* Significant visual/auditory problem.
* Botox injection and/or surgery of the upper limb in the past 12 months.
* Fixed deformities in the affected upper extremity.

Ages: 4 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: Participants will be recruited from the Outpatient Clinic of Faculty of Physical Therapy, Cairo University, Abo El-reesh Hospital and the Outpatient Clinic of Al-Minya General Hospital, Al-Minya Governorate.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Test of Arm Selective Control | 1/2/2021 to 30/4/2021
  The goal of the assessment is to systematically evaluate a person's ability to move the upper extremity with selective voluntary motor control by observing movement control, coordination, fluency, mirroring, and speed at each joint, and then assigning a grade. Each joint is scored as a 0, 1, or 2. The joints of the affected limb are summed for a limb score for a total score. The maximum score is 16 per side, or 32 points in total (in hemiplegia assess the affected side only) with higher score indicates better performance. Admiration of the teat items and scoring will be conducted according to the scale user instructions.

SECONDARY OUTCOMES:
Hand Held Dynamometer | 1/2/2021 to 30/4/2021
  to evaluate hand grip strength
Quality of Upper Extremity Skill Test | 1/2/2021 to 30/4/2021
  to assess upper limb function

CONTACTS AND LOCATIONS:
Overall Officials: Maya Galal, Phd, Study Director — Cairo University; Radwa Gomaa, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt